CLINICAL TRIAL: NCT00372333
Title: A Multiple-Dose, Open-Label Safety, Compliance, and Usage Evaluation Study of Epicutaneously Applied IDEA-033 in Joint / Musculoskeletal Pain or Soft Tissue Inflammation
Brief Title: IDEA-033 Open Label Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IDEA AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-033-III-01
Record Dates: First submitted 2006-09-04; First posted 2006-09-06 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Joint Pain; Musculoskeletal Pain; Stiffness; Soft Tissue Inflammation in Designated Target Area(s)
Keywords: musculoskeletal pain; soft tissue inflammation; IDEA-033
MeSH Terms: conditions — Arthralgia; Musculoskeletal Pain

INTERVENTIONS:
Drug: IDEA-033

SUMMARY:
The main aim of the study is to evaluate safety, efficacy, compliance, and usage of epicutaneously applied IDEA-033 in joint / musculoskeletal pain or soft tissue inflammation.

DETAILED DESCRIPTION:
Multi-centre, one arm, multiple dose, open-label, at home usage study. Adult volunteers experiencing joint pain, musculoskeletal pain, stiffness, or soft tissue inflammation will be screened for study participation.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years or older
* agree to refrain from chronic usage of NSAIDs or any other analgesics or anti-inflammatory drugs other than those provided during the course of the study or documented sporadic concomitant analgesics
* joint pain, musculoskeletal pain, stiffness, or soft tissue inflammation in designated target area(s) that are appropriate for self-treatment with a topical analgesic or where availability of a second person can be guaranteed in case self-treatment is not possible
* healthy skin in the target area(s)

Exclusion Criteria:

* known hypersensitivity to IDEA-033 or other NSAIDs
* history of coagulation disorders
* history of peptic ulcers or gastric intolerance with NSAIDs
* urinary tract infection
* clinically significant renal, hepatic, or gastric disease
* acute or chronic coexisting illness qualifying for exclusion according to clinical judgement of the investigator
* clinical laboratory values outside normal range deemed clinically significant by the investigator
* Narcotics-containing products within 7 days of administering IMP
* Malignancy within the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
description of AE profile
changes in laboratory values
IDEA-033 plasma levels
visual assessment of skin at target area(s)
physical exam
vital signs

SECONDARY OUTCOMES:
evaluation of efficacy by real time feedback

CONTACTS AND LOCATIONS:
Overall Officials: Ilka Rother, Principal Investigator — X-pert-med GmbH Munich
Locations (1):
- X-pert med GmbH / Ilka Rother, Gräfelfing, Bavaria, Germany